

## **CONSENT FORM**

"Comparative evaluation of impact of sodium hypochlorite on physical properties of finishing ProTaper Gold and Dia-X ProTaper Files: An In vitro Randomized control trial study."

Principle Investigator: Dr. Iqra Kamal 15-March-2021



## **CONSENT FORM**

Research Title: "Comparative evaluation of impact of sodium hypochlorite on physical properties of finishing ProTaper Gold and Dia-X ProTaper Files: An In vitro Randomized control trial study."

Principal Investigator: Dr. Iqra kamal

You are requested to participate in a research study described below. Please read the consent form thoroughly. Please note that your participation in this study is completely on voluntary basis.

<u>Purpose of this study:</u> This study will aid in providing a better quality of root canal treatment.

<u>Participation:</u> You are being requested to voluntarily donate your extracted tooth for research purpose.

<u>Confidentiality:</u> All information regarding your identity will be kept confidential.

<u>Possible Risks and Benefits:</u> There are no associated risks nor will you receive any financial benefit from participation in this study.

## **CONSENT:**

| I have thoroughly read and understood this consent form. I understand that my |
|---|
| participation in this study is voluntary. I hereby give my consent to participate in this |
| study. |

| Participant`s Signature: | Date: |
|--------------------------|-------|
| 1 0 | |